CLINICAL TRIAL: NCT03310489
Title: Digitalized Cognitive-behavioral Intervention for Anxiety Among School Children. A Randomized Controlled Study
Brief Title: A Randomized Controlled Study of Digitalized Cognitive-behavioral Intervention for Childhood Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Andre Sourander, Professor (child psychiatry), University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANXIETY-2017
Record Dates: First submitted 2017-09-30; First posted 2017-10-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitalized cognitive-behavioral intervention (Experimental)
  Interventions: Behavioral: Digitalized cognitive-behavioral intervention for anxiety
- Psychoeducation about anxiety (Active Comparator)
  Interventions: Behavioral: Psychoeducation about anxiety

INTERVENTIONS:
Behavioral: Digitalized cognitive-behavioral intervention for anxiety — An internet-based CBT, including telephone coaching
  Arms: Digitalized cognitive-behavioral intervention
Behavioral: Psychoeducation about anxiety — Psychoeducative material about anxiety in internet
  Arms: Psychoeducation about anxiety

SUMMARY:
The aim of the study is to evaluate the effectiveness of a digitalized cognitive-behavioral treatment for anxiety among school aged children. The participants are screened from the general population, as a part of the routine school health care check-ups. Half of the children with anxiety will receive the digitalized treatment program, while the other half will receive education about anxiety in internet.

ELIGIBILITY:
Inclusion Criteria:

- Scoring ≥22 on SCARED

Exclusion Criteria:

* no access to internet
* insufficient language (Finnish until summer 2019, Finnish and Swedish from autumn 2019 onwards, when also Swedish version of the intervention was available) skills
* visual or hearing impairment that hinders the use of the program
* the child's mental retardation, autism spectrum disorder, suicidal intentions or severe mental disorder
* the child's psychotherapy (ongoing or starting within 6 months)
* the child's medication (for anxiety) started / changed within 2 months
* current involvement with child protection services (i.e., removal of child custody, investigation of child abuse or neglect)
* parent's severe psychiatric / somatic disease or other reason that hinders the parent to actively participate in the program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 6 months follow up; the Screen for Child Anxiety Related Disorders - child and parent reports | Change from baseline to 6 months follow up; symptoms during the last three months
  Comprises of 41 items assessing symptoms of general anxiety, separation anxiety, panic disorder, social anxiety, and school phobia; scoring 0-82 (higher score meaning more symptoms)

SECONDARY OUTCOMES:
Change from Baseline to 6 months follow up; the Child Anxiety Impact Scale - child and parent reports | Change from baseline to 6 months follow up; impact of anxiety during the last month
  Comprises of 27 items assessing the impact of anxiety on the daily life of the children at home, school and with friends; scoring 0-81 (higher score meaning higher impact of anxiety)
Change from Baseline to 6 months follow up (in the Intervention group); the Development and Well-Being Assessment - child and parent reports | Change from baseline to 6 months follow up; varying time windows for different diagnoses
  A diagnostic interview to assess anxiety disorders among 2-17-year-old children
Change from Baseline to 6 months follow up; the Revised Children Quality of Life - Questionnaire - child and parent reports | Change from baseline to 6 months follow up; QoL during the last week
  Comprises of 24 items assessing the health-related quality of life divided into six subscales: physical, psychological, self-esteem, family, social life, and school; scoring 24-96 (higher score meaning higher QoL)
Change from Baseline to 6 months follow up; the Child Depression inventory - child report | Change from baseline to 6 months follow up; symptoms during the last two weeks
  Comprises of 28 items assessing the child's depressive symptoms; scoring 0-54 (higher score meaning more symptoms)
Change from Baseline to 6 months follow up; the Strengths and Difficulties Questionnaire, extended version - parent report | Change from baseline to 6 months follow up; symptoms during the last six months
  Comprises of 25 items assessing the child's psychiatric symptoms and positive attributes, and an impact supplement; scoring 0-40 (prosocial scale is not included in the total score) (higher score meaning more problems)
Change from Baseline to 6 months follow up of the relations with peers and school (not a standardized scale) | Change from baseline to 6 months follow up
  Experience of being bullied (traditional and cyberbullying), and feelings about school and teachers
Change from Baseline to 6 months follow up; the Brief resilience scale - parent report (parental resilience) | Change from baseline to 6 months follow up; experience of the current resilience
  Comprises of six items assessing resilience; scoring 6-36 (higher score meaning higher resilience)
Change from Baseline to 6 months follow up; the Depression Anxiety and Stress Scale Short Form - parent report (parental depression, anxiety and stress) | Change from baseline to 6 months follow up; symptoms during the last week
  Comprises of 21 items assessing parental depression, anxiety and stress; scoring 0-63 (higher score meaning more symptoms)
Change from Baseline to 6 months follow up; the Customised Client Receipt Inventory Questionnaire - parent report | Change from baseline to 6 months follow up; service use during the last six months
  Assesses the child's use of school support services, and social and health care services

CONTACTS AND LOCATIONS:
Locations (1):
- Child Psychiatric Research Center, University of Turku, Turku, Finland

REFERENCES:
- [Derived] Sourander A, Korpilahti-Leino T, Kaajalaakso K, Ristkari T, Hinkka-Yli-Salomaki S, Stahlberg T, Luntamo T. Internet-Based Cognitive-Behavioral Therapy Intervention Master Your Worries With Telephone Coaching for Anxious Finnish Children Aged 10-13 Years: A Population-Based Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2025 Nov;64(11):1281-1294. doi: 10.1016/j.jaac.2024.11.024. Epub 2025 Feb 4. PMID 39914585
- [Derived] Luntamo T, Korpilahti-Leino T, Ristkari T, Hinkka-Yli-Salomaki S, Kurki M, Sinokki A, Lamminen K, Saanakorpi K, Saarinen S, Maunuksela M, Sourander S, Toivonen K, Zadkova A, Suilamo M, Casagrande L, Palmroth J, Sourander A. Internet-assisted cognitive behavioural therapy with telephone coaching for anxious Finnish children aged 10-13 years: study protocol for a randomised controlled trial. BMJ Open. 2021 Jun 23;11(6):e045474. doi: 10.1136/bmjopen-2020-045474. PMID 34162641